CLINICAL TRIAL: NCT03173001
Title: Intestinal Helminths and Protozoan Infections in Patients With Colorectal Cancer: Prevalence and Possible Association With Cancer Pathogenesis
Brief Title: Possible Association of Intestinal Helminths and Protozoa With Colorectal Cancer Pathogenesis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Research Institute of Epidemiology, Microbiology and Infectious Diseases, Uzbekistan (Other Government)
Responsible Party: Principal Investigator, Svetlana Osipova, MD, PhD, DS, Professor, Research Institute of Epidemiology, Microbiology and Infectious Diseases, Uzbekistan
Other Study IDs: ADCC 15 21 2
Record Dates: First submitted 2017-05-29; First posted 2017-06-01 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Cancer; Colorectal Cancer Metastatic; Intestinal Parasite; Protozoan Infections
Keywords: intestinal helminths; protozoan infections;; colorectal cancer; chemotherapy; cancer pathogenesis;
MeSH Terms: conditions — Colorectal Neoplasms; Intestinal Diseases, Parasitic; Protozoan Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Patients with colorectal cancer: Patients hospitalized with colorectal cancer at the Department of Coloproctology of Republican Oncology Research Center.
  Interventions: Diagnostic Test: Parasitological examination
- Population: The control group includes residents of Tashkent city without any complaints from gastrointestinal tract matched by gender and age to the patients with colorectal cancer.
  Interventions: Diagnostic Test: Parasitological examination
- Patients with CRC without metastases: Patients hospitalized with colorectal cancer at the Department of Coloproctology of Republican Oncology Research Center.
  Interventions: Diagnostic Test: Parasitological examination
- Patients with CRC with metastases: Patients hospitalized with colorectal cancer at the Department of Coloproctology of Republican Oncology Research Center.
  Interventions: Diagnostic Test: Parasitological examination
- Patients with CRC before operation: Patients hospitalized with colorectal cancer before operation at the Department of Coloproctology of Republican Oncology Research Center.
  Interventions: Diagnostic Test: Parasitological examination
- Patients with CRC after operation: Patients hospitalized with colorectal cancer after operation at the Department of Coloproctology of Republican Oncology Research Center.
  Interventions: Diagnostic Test: Parasitological examination
- Patients with CRC before chemotherapy: Patients hospitalized with colorectal cancer before operation and chemotherapy at the Department of Chemotherapy of Republican Oncology Research Center.
  Interventions: Diagnostic Test: Parasitological examination
- Patients with CRC after chemotherapy: Patients hospitalized with colorectal cancer after operation and chemotherapy at the Department of Chemotherapy of Republican Oncology Research Center.
  Interventions: Diagnostic Test: Parasitological examination

INTERVENTIONS:
Diagnostic Test: Parasitological examination — Three stool samples for parasitological examination will be taken from control subjects and CRC patients at 1-2 days interval.
  Other Names: Coproscopy

SUMMARY:
Colorectal cancer (CRC) has the third highest cancer incidence in the world. There is mounting evidence that the intestinal microbiota plays an important role in colorectal carcinogenesis. but there is no information on protozoa of intestinal microbiota except Blastocystis hominis, although data on this issue is scarce. In this study we are going to evaluate the prevalence of intestinal helminthes and protozoa in CRC patients and control group that includes random residents. Patients will be examined before, after surgery and chemotherapy. Parasites and protozoan infection intensity will be estimated by triple coproscopy.

DETAILED DESCRIPTION:
The study will be conducted on the basis of Research Institute of Epidemiology, Microbiology and Infectious Diseases and Research Center of Oncology, Ministry of Public Health of the Republic of Uzbekistan.

All the CRC patients from Research Center of Oncology will be examined with their written concent. Diagnosis of CRC is based on the results of clinical examination, endoscopic, histological, X-ray and laboratory data according to International Classification proposed by the American Joint Committee on Cancer (AJCC) with application TNM (T-tumor, N-nodus, M-metastases) for diagnosis. Descriptors in T (primary tumor) mean the degree of the tumor spreading in layers of the intestine; descriptors in N mean absence of metastases or the number of lymph nodes with metastases; descriptors in M shows absence or presence of remote metastases.

The control group will be a random residents of Tashkent city without any complaints from gastrointestinal tract matched by gender and age to the patients with CRC. Age of individuals under examination will be taken at the range from 17 to 90 years old.

Collection of stool samples Three stool samples for parasitological examination will be taken from both control subjects and CRC patients at 1-2 days interval. Stool samples were collected in individual containers, containing 5 ml of Turdiev's preservative provided conservation and staining of protozoa cysts and eggs of worms for a year. The Turdiev's preservative includes:80 ml of 0.2% aqueous solution of sodium nitrite, 10 ml of formaldehyde, 2 ml of glycerin, 8 ml of Lugol's solution, 250 ml of distilled water.

Collection of material for C. parvum (Cryptosporidium parvum) detection in stool samples will be carried out by preparation of fresh feces thin smears.

Stool samples examination Parasitological diagnosis will be performed by triple coproscopy using formalin - ethyl acetate concentration technique. For preparations staining Lugol's solution was used. The intensity of protozoa will be estimated by the number of protozoa in the field of view (ocular x10, objective x40), the number of protozoa will be calculated at least in 10 fields of view. 1-2, 3-4 and 5-6 microorganisms in a field of view were considered as infection of low, mean and high intensity respectively.

Modified Ziehl- Neelsen method will be used for staining and detection of C. parvum preparations. The stained smears will be observed with ×100 oil immersion lens for the presence of C. parvum.

Parasitological examination of the additional group of the patients obtained chemotherapy will be carried out before and after surgery and complete course of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* All patients with colorectal cancer before, after surgery and chemotherapy.

For control group:

* Includes all individuals that doesn't have any complaints from gastrointestinal tract

Exclusion Criteria:

* Age before 18.
* Patients with other gastrointestinal disorders
* Patients with any chronic concomitant diseases

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with colorectal cancer hospitalized in Department of Coloproctology at Research Center of Oncology. Diagnosis of colorectal cancer is based on the results of clinical examination, endoscopic, histological, X-ray and laboratory data according to International Classification proposed by the American Joint Committee on Cancer (AJCC) with application TNM for diagnosis.
  The control group will be a residents of Tashkent city without any complaints from gastrointestinal tract matched by gender and age to the patients with CRC.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of intestinal helminths in patients with colorectal cancer and association with cancerogenesis | from 2015 to 2018 years
  In this study we expect to find intestinal helminths in patients with colorectal cancer and determine their role in the development of colorectal cancer
Prevalence of Lamblia intestinalis and Cryptosporidium parvum in patients with colorectal cancer and association with cancerogenesis | from 2015 to 2018 years
  In this study we expect to find pathogenic protozoa in patients with colorectal cancer and determine their role in the development of colorectal cancer
Prevalence of intestinal protozoa (commensals) in patients with colorectal cancer and association with cancerogenesis | from 2015 to 2018 years
  In this study we are going to determine their prevalence and role in the development of colorectal cancer

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Toychiev A, Abdujapparov S, Imamov A, Navruzov B, Davis N, Badalova N, Osipova S. Intestinal helminths and protozoan infections in patients with colorectal cancer: prevalence and possible association with cancer pathogenesis. Parasitol Res. 2018 Dec;117(12):3715-3723. doi: 10.1007/s00436-018-6070-9. Epub 2018 Sep 15. PMID 30220046